CLINICAL TRIAL: NCT07180095
Title: Intranasal Dexmedetomidine Versus Intranasal Ketamine for Preoperative Sedation in Pediatrics
Brief Title: Children of Age 2-6years Undergoing Elective Surgery Will be Divided Into Two Groups Randomly. This Study Aims to Evaluate if Intranasal Dexmedetomidine is Better Than Intranasal Ketamine in Producing Sedation and Reducing Parent Separation Anxiety Before Surgery.
Acronym: DREAM-Kids
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Aimon Irshad, Principal Investigator, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: aimusa00
Record Dates: First submitted 2025-09-04; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Sedation; Preoperative Anxiety Experienced by the Pediatric Patient; Anxiolytic Effect; Sedation and Analgesia
Keywords: Preoperative Sedation; Hemodynamic changes; Dexmedetomidine; Dexmedetomidine vs Ketamine
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal Dexmedetomidine (Active Comparator): Received Intranasal Dexmedetomidine
  Interventions: Drug: Intranasal dexmedetomidine
- Intranasal ketamine (Experimental): Received Intranasal Ketamine.
  Interventions: Drug: Intranasal ketamine

INTERVENTIONS:
Drug: Intranasal dexmedetomidine — intranasal dexmedetomidine 2mcg/kg
  Arms: Intranasal Dexmedetomidine
Drug: Intranasal ketamine — intranasal ketamine 2mg/kg
  Arms: Intranasal ketamine

SUMMARY:
This study aims to compare intranasal dexmedetomidine versus intranasal ketamine as a premedication in children undergoing surgery in our population. Hypothesis is Intranal dexmedetomidine is better than intranasal ketamine in producing preoperative sedation in pediatric patients undergoing surgery under general anesthesia.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, controlled trial with Minimum 6 months of data collection. Patients will be randomly divided into 2 groups; Group D and Group K with 30 patients in each group. Group D will receive dexmedetomidine 2 mcg/kg intranasal, diluted in normal saline to a total volume of 1 mL and will be administered 0.5 mL per nostril while group K will receive ketamine 2mg/kg intranasal, diluted in normal saline to a total volume of 1 mL similarly divided into two nostrils. The study drugs will be prepared by a second anesthesiologist who will not be involved in subsequent assessments. The calculated dose for each patient will be administered 30 minutes before induction of anesthesia in preoperative holding area in parental/guardian presence. Sedation level will be assessed at 10 minutes interval for the next 30 minutes or until the child will be shifted to the operating room using MOAA/S and ease of parental separation will be scored using PSAS. All patients will be monitored using standard ASA monitoring (ECG, non-invasive blood pressure , pulse oximetry) before induction then every 5 minutes till the end of surgery or a maximum of 1 hour in the operating room. All patients will be induced with 6-8% sevoflurane in 100% oxygen and a 24-G IV access will be secured once the child is asleep. Nalbuphine 0.1 mg/kg IV, atracurium 0.5mg/kg IV (or rocuronium 0.6mg/kg if there's contraindication to atracurium). After endotracheal intubation or laryngeal mask airway (LMA) insertion, all patients will be maintained with 50% O2 in air with isoflurane. Ventilation will be adjusted to maintain an end tidal CO2 concentration between 30-40mmHg. All patients will be given IV paracetamol 20mg/kg as part of multimodal analgesia. If heart rate drops <70 bpm, atropine 10mcg/kg I/V will be used and hypotension will be treated with IV adrenaline 10mcg/kg. Neuromuscular blockade will be reversed with 50mcg/kg neostigmine and 10mcg/kg glycopyrolate. After regaining regular and spontaneous breathing, the endotracheal tube or LMA will be removed and the child will be shifted to post-anesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* American society of Anesthesiologist (ASA) class-I and II
* Children 2-6 years of age undergoing elective surgery

Exclusion Criteria:

* Known hypersensitivity to study drugs
* Refusal of consent
* Known renal, hepatic or cardiac dysfunction
* Nasal deformity or pathology
* Recent upper respiratory infection (within 2 weeks)
* Children undergoing neurosurgery or ophthalmic surgery

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Sedation score as assessed by MOAA/S | 6 months
  Modified Observer's Assessment of Alertness/ Sedation scale (MOAA/S):
  6 = Appears alert and awake, responds readily to name spoken in a normal tone 5 = Appears asleep but responds readily to name spoken in a normal tone 4 = Lethargic response to name spoken in a normal tone 3 = Responds only after the name is called loudly or repeatedly 2 = Responds only after mild prodding or shaking
  1 = Does not respond to mild prodding or shaking

SECONDARY OUTCOMES:
Ease of parental separation using PSAS | 6 months
  Parental Separation Anxiety Score (PSAS):
  1. = Excellent (unafraid, cooperative)
  2. = Good (slight fear or crying, easily reassured)
  3. = Fair (moderate fear, not quiet with reassurance)
  4. = Poor (crying, needing restraint)
Incidence of hypotension and bradycardia in the two groups | 6 months
  Intraoperative hypotension and bradycardia will be monitored before induction then every 5 minutes till the end of surgery or a maximum of 1 hour in the operating room.